CLINICAL TRIAL: NCT01223729
Title: Acetyl-L-Carnitine Reduces Depression and Improves Quality of Life in Patients With Minimal Hepatic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Mariano Malaguarnera, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8-12-00 A
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2000-12

CONDITIONS: Minimal Hepatic Encephalopathy
Keywords: Acetyl-L-carnitine;; Minimal hepatic encephalopathy;; Quality of life;; Depression.
MeSH Terms: conditions — Depression | interventions — Acetylcarnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetyl-L-Carnitine (Experimental)
  Interventions: Drug: Acetyl-L-Carnitine
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Acetyl-L-Carnitine — 2 g acetyl-L carnitine twice a day
  Arms: Acetyl-L-Carnitine
Other: placebo — placebo twice per day
  Arms: placebo

SUMMARY:
Minimal hepatic encephalopathy represents a common complication present in well-compensated cirrhotic patients that impairs patients daily functioning and health-related quality of life. Acetyl-L-carnitine has been shown to be useful in improving blood ammonia and cognitive functions in cirrhotic patients with minimal hepatic encephalopathy. This study evaluated the effects of acetyl-L-carnitine treatment on health related quality of life and on depression in patients with minimal hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed as having cirrhosis at the outpatient Internal Medicine of the Department of Senescence of Cannizzaro Hospital (Catania) were candidates for enrolment. The diagnosis of cirrhosis was based on clinical, biochemical and ultrasonographic or liver histological data.

Exclusion Criteria:

* Exclusion criteria were overt hepatic encephalopathy or a history of overt HE; history of recent alcohol intake; infection; recent antibiotic use or gastrointestinal bleeding; history of recent use of drugs affecting psychometric performances like benzodiazepines, antiepileptics or psychotropic drugs; a history of shunt surgery or transjugular intrahepatic portosystemic shunt for portal hypertension; electrolyte imbalance; renal impairment; hepatocellular carcinoma; severe medical problems such as congestive heart failure, pulmonary disease or neurological or psychiatric disorder that could influence quality of life measurement; inability to perform neuropsycological tests.

Ages: 34 Years to 67 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 67
Dates: Start 2002-04; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- Cannizzaro Hospital, Catania, Italy

REFERENCES:
- [Background] Malaguarnera M, Gargante MP, Cristaldi E, Vacante M, Risino C, Cammalleri L, Pennisi G, Rampello L. Acetyl-L-carnitine treatment in minimal hepatic encephalopathy. Dig Dis Sci. 2008 Nov;53(11):3018-25. doi: 10.1007/s10620-008-0238-6. Epub 2008 Mar 21. PMID 18357530